CLINICAL TRIAL: NCT00515294
Title: Acute and Residual Effects of Beer VS. Caffeinated Beer On Simulated Driving
Brief Title: Acute and Residual Effects of Caffeinated Beer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Brown University (Other); University of Michigan (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: H-26002; R49CE000946 (NIH)
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Neurobehavioral Manifestations; Drug Related Sleep Disturbance; Alcohol Intoxication
Keywords: Caffeine; Alcohol; Alcohol Consumption; Residual Effects; Family History; Psychomotor Vigilance Test; Driving Simulation; Reaction Time
MeSH Terms: conditions — Neurobehavioral Manifestations; Alcoholic Intoxication; Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1Caffeinated Alcoholic Beer (Experimental): Caffeinated Alcoholic beer
  Interventions: Drug: Caffeinated Alcoholic Beer
- 2Non-Caffeinated Alcoholic Beer (Active Comparator): Non-Caffeinated Alcoholic beer
  Interventions: Other: Non-Caffeinated Alcoholic Beer
- 3Caffeinated Non-Alcoholic Beer (Active Comparator): Caffeinated Non-Alcoholic Beer
  Interventions: Drug: Caffeinated Non-Alcoholic Beer
- 4Non-Caffeinated, Non-Alcoholic Beer (Placebo Comparator): Non-Caffeinated, Non-Alcoholic Beer
  Interventions: Other: Non-Caffeinated, Non-Alcoholic Beer

INTERVENTIONS:
Drug: Caffeinated Alcoholic Beer — Alcoholic Beer plus Caffeine Citrate powder.
  Other Names: 69mg caffeine/12oz glass of regular beer
  Arms: 1Caffeinated Alcoholic Beer
Other: Non-Caffeinated Alcoholic Beer — Alcoholic Non-Caffeinated Beer
  Arms: 2Non-Caffeinated Alcoholic Beer
Drug: Caffeinated Non-Alcoholic Beer — Non-Alcoholic Beer plus Caffeine Citrate powder.
  Other Names: 69mg caffeine/12oz glass of non-alcoholic beer
  Arms: 3Caffeinated Non-Alcoholic Beer
Other: Non-Caffeinated, Non-Alcoholic Beer — Non-Alcoholic Beer
  Other Names: Placebo
  Arms: 4Non-Caffeinated, Non-Alcoholic Beer

SUMMARY:
The aim of this study is to develop information about the acute and residual effects of a new product being targeted to young adults. Using a double placebo-controlled 2 X 2 factorial model study design, we will compare the acute and residual effects on driving impairment of caffeinated alcohol, non-caffeinated alcohol, caffeinated placebo, and non-caffeinated placebo. Under the alcohol conditions, participants will receive sufficient alcoholic beverage to attain a blood alcohol concentration (BAC) of .12 g%. Participants will be 144 undergraduate and graduate students, and recent college graduates.

DETAILED DESCRIPTION:
Caffeinated alcoholic beverages target young adults with the promise that the caffeine will counteract the sedating effects of alcohol and thus let the consumer remain alert and active longer, while continuing to drink. It is likely that in the minds of some young people, this promise also translates into the idea that mixing caffeine with alcohol allows one to drive more safely than would be possible after having consumed an equivalent amount of non-caffeinated alcoholic beverage. These are dangerous assumptions because (1) alertness may not indicate the absence of impairment under intoxication and (2) next-day impairment from the residual effects of heavy drinking may be exacerbated by mixing caffeine and alcohol. We will compare the acute and residual effects of caffeinated and non-caffeinated beer in terms of a highly relevant outcome - the ability to drive safely.

The long-term objectives of this program of research are to investigate factors that predict or contribute to performance decrements after alcohol ingestion, with a focus on behaviors most relevant to public health, such as driving. The primary specific aims of the proposed work are:

AIM 1: To compare the acute effects of caffeinated alcohol, non-caffeinated alcohol, caffeinated placebo, and non-caffeinated placebo on driving-related impairment, as measured by performance on a driving simulator and the Psychomotor Vigilance Test (PVT), a test of sustained attention/reaction time. We hypothesize that caffeinated beverage will result in less impaired simulated driving ability and better PVT performance acutely, compared to non-caffeinated beverage, but that performance on these measures following both caffeinated and non-caffeinated beverage be impaired relative to placebo beverages.

AIM 2: To compare the residual effects of caffeinated alcohol, non-caffeinated alcohol, caffeinated placebo, and non-caffeinated placebo on next-day driving-related impairment, as measured by a driving simulator and the PVT. We hypothesize that caffeinated beverage will result in greater impairment in next-day simulated driving and attention/reaction time, relative to non-caffeinated beverage, and that performance following both caffeinated and non-caffeinated alcoholic beverages will be impaired relative to corresponding placebo beverages.

AIM 3: To compare the acute effects of caffeinated alcohol, non-caffeinated alcohol, caffeinated placebo, and non-caffeinated placebo on self-rated ability to drive, as measured by a self assessment of ability-to-drive questionnaire, and estimate of blood alcohol concentration (BAC). We hypothesize that caffeinated alcoholic beverages will result in greater confidence in ability to drive and lower estimates of BAC, compared to non-caffeinated alcoholic beverages, but that for both alcoholic beverages, confidence in driving ability will be lower and estimates of BAC will be greater, relative to placebos.

AIM 4: To compare the residual effects of caffeinated alcohol, non-caffeinated alcohol, caffeinated placebo, and non-caffeinated placebo on self-rated ability to drive. We hypothesize that caffeinated alcoholic beverage will result in lower confidence in ability to drive and higher estimates of BAC, compared to non-caffeinated alcoholic beverage, but that for both alcoholic beverages, confidence in driving ability will be lower and estimates of BAC will be greater, relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* College students, graduate students, or recent graduates
* Between the ages of 21 and 30 years inclusive (as verified by valid drivers license)
* Who, if a student, reports good academic standing
* Have not been diagnosed with a sleep disorder
* Are not daily smokers
* At least occasionally in the past month, consume five drinks (for men) or more (four or more if female [based on Flannery et al 2002]) during a single drinking episode
* Have a valid drivers license, so as to include only people who know how to drive.

Exclusion Criteria:

* Scores of 5 or more on a screening measure for alcoholism (the short version of the Michigan Alcohol Screening Test [SMAST])
* A history of counseling or treatment for chronic substance abuse by self-report
* Daily smoker (to mitigate confounding of caffeine by nicotine withdrawal, or acute nicotine administration, smokers will be excluded from participation)
* Current use of medications that affect the sleep/wake cycle or daytime alertness or that are contraindicated for alcohol
* Presence of a health condition that contraindicates alcohol
* Diagnosis of a sleep disorder (sleep apnea, narcolepsy, periodic limb movement, restless legs syndrome, circadian rhythm disorder, and insomnia)
* Use of recreational drugs (e.g., marijuana) while participating in the study
* Working overnight shifts
* Female and pregnant, nursing, or not using reliable birth control
* Participants who have traveled across two or more time zones in the last month will be rescheduled for later participation (minimum of 1 month from time-zone travel)
* On average consume greater than 4 cups of coffee per day (>400 mg/day)
* Participants who report ever getting motion sick during screening or become motion sick after practicing on the driving simulator during Session 1.
* Weigh more than 230 Lbs.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Howland, PhD, MPH, Principal Investigator — Boston University
Locations (1):
- General Clinical Research Center, Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howland J, Rohsenow DJ, Arnedt JT, Bliss CA, Hunt SK, Calise TV, Heeren T, Winter M, Littlefield C, Gottlieb DJ. The acute effects of caffeinated versus non-caffeinated alcoholic beverage on driving performance and attention/reaction time. Addiction. 2011 Feb;106(2):335-41. doi: 10.1111/j.1360-0443.2010.03219.x. Epub 2010 Dec 6. PMID 21134017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited via newspaper ads and social media.
Groups:
- 4Non-Alcoholic, Non-Caffeinated Beer: Non-Caffeinated, Non-Alcoholic Beer: Non-Alcoholic Beer
Period: Overall Study
Arm/Group | 1Caffeinated Alcoholic Beer | 2Non-Caffeinated Alcoholic Beer | 3Caffeinated Non-Alcoholic Beer | 4Non-Alcoholic, Non-Caffeinated Beer
Started | 38 | 39 | 38 | 39
Completed | 29 | 36 | 27 | 35
Not Completed | 9 | 3 | 11 | 4
Not completed — Lost to Follow-up | 3 | 2 | 3 | 1
Not completed — Driver simulator problems | 1 | 1 | 1 | 3
Not completed — Caffeine amount inaccurate | 5 | 0 | 7 | 0

BASELINE CHARACTERISTICS:
Population: We compared participants across groups by age and sex.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1Caffeinated Alcoholic Beer | 2Non-Caffeinated Alcoholic Beer | 3Caffeinated Non-Alcoholic Beer | 4Non-Alcoholic, Non-Caffeinated Beer | Total
Number analyzed (Participants) | 29 | 36 | 27 | 35 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 36 | 27 | 35 | 127
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 13 | 16 | 60
  Male | 15 | 19 | 14 | 19 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 3 | 5 | 3 | 5 | 16
  Race: Black/African American | 1 | 2 | 0 | 1 | 4
  Race: White | 22 | 27 | 20 | 26 | 95
  Race: More than one race | 0 | 1 | 2 | 2 | 5
  Race: Unknown, not reported | 3 | 1 | 2 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 29 | 36 | 27 | 35 | 127

OUTCOME MEASURES:

1. Primary Outcome: Lane Position Deviation
Description: The reported lane position deviation indicates the position of the car relative to the center line in feet in the driver simulator. A deviation of 0 indicates no deviation from the center line (the car is positioned farthest from the road edge). Negative numbers indicate deviations to the right of the center line with the car positioned within the lane closer to the road edge. Positive numbers indicate deviations to the left of the center line with the car positioned in the lane of oncoming traffic closer to the road edge
Time Frame: 30 minutes post dosing
Population: Driver simulator did not work properly for 6 participants. Their data are not included.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | 1Caffeinated Alcoholic Beer | 2Non-Caffeinated Alcoholic Beer | 3Caffeinated Non-Alcoholic Beer | 4Non-Alcoholic, Non-Caffeinated Beer
Number analyzed (Participants) | 28 | 35 | 26 | 32
feet | -1.25 (.61) | -1.36 (.85) | -1.22 (.53) | -1.21 (.77)

2. Secondary Outcome: Psycho-motor Vigilance Test (PVT)
Description: Participants completed 10 test trials to assess their psycho-motor response using a hand held box that randomly starts a scroll of numbers in milliseconds and as soon as it starts to scroll the participant needs to press a button to stop the scrolling. The mean and standard deviations for the 10 tests were calculated as a single outcome score for each study arm. Response times were measured in milliseconds. The lower the number of milliseconds the faster the response to the random stimuli.
Time Frame: 30 minutes post dosing
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | 1Caffeinated Alcoholic Beer | 2Non-Caffeinated Alcoholic Beer | 3Caffeinated Non-Alcoholic Beer | 4Non-Alcoholic, Non-Caffeinated Beer
Number analyzed (Participants) | 29 | 36 | 27 | 35
milliseconds | 278.7 (46.6) | 293.3 (47.0) | 233.1 (22.3) | 241.8 (25.6)

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- 1Caffeinated Alcohol: Caffeinated Alcoholic Beer: Alcoholic Beer plus Caffeine Citrate powder.
- 2Non-Caffeinated Alcohol: Non-Caffeinated Alcoholic Beer: Alcoholic Non-Caffeinated Beer
Arm/Group | 1Caffeinated Alcohol | 2Non-Caffeinated Alcohol | 3Caffeinated Non-Alcoholic Beer | 4Non-Alcoholic, Non-Caffeinated Beer
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/36 | 0/27 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/36 | 0/27 | 0/35
Other Adverse Events (participants affected / at risk) | 0/29 | 0/36 | 0/27 | 0/35

LIMITATIONS AND CAVEATS:
Difficulties with the driver simulator resulted in invalid data for 6 participants so their results were not included in the lane position deviation results. Inaccurate caffeine doses resulted in exclusion of 12 participants from the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No